CLINICAL TRIAL: NCT06405815
Title: Development of a Tumor and Peritumor Radiomics-based Model to Predict the High-risk Surgical Margin and Prognosis of T3 and T4 Non-Small Cell Lung Cancer
Brief Title: A Radiomic Model for Risk of Local Recurrence and DFS for T3 and T4 Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Guangming Lu, Director of the Medical Imaging Center of the Jinling Hospital, Jinling Hospital, China
Other Study IDs: JinlingHospital_lungcancer
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: non-small cell lung cancer; surgical margin; DFS; radiomics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Margins of Excision | interventions — Tumor Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- high-risk surgical margin: High-risk margins were defined as R1 or R2 surgical margins or local recurrence during follow-up.
  Interventions: Other: tumor and peritumor radiomic feature
- Low-risk surgical margin: Low-risk margins were defined as R0 surgical margin meanwhile arising distant metastasis during follow-up.
  Interventions: Other: tumor and peritumor radiomic feature

INTERVENTIONS:
Other: tumor and peritumor radiomic feature — extracted the tumor and peritumor radiomic feature from the preoperative enhanced chest CT

SUMMARY:
The investigators retrospectively collected the participants with T3 and T4, N0-2, M0 NSCLC patients resected between January 2013 to December 2021 for training and internal validation. The Clinical data, preoperative laboratory results and images were collected. High-risk margins were defined as R1 or R2 surgical margins or local recurrence during follow-up, and the investigators also collected the disease-free survival time. On the Deepwise multi-modal research platform, the images were semi-automatically segmented and expanded outward by 3mm to obtain the peritumor tissue. PyRadiomics was used to extract the radiomic features. LASSO was used to select the features and tumor radiomics model, peritumor model and combined model were built using 5-fold cross-validation. And it was further tested on the independent cohort. Discrimination was assessed by using the C-index and area under the receiver operating characteristic curve (AUC), sensibility, specificity.

ELIGIBILITY:
Inclusion Criteria:

* patients with T3 and T4 stage NSCLC；
* available preoperative chest CTE within two weeks of surgery

Exclusion Criteria:

* inadequate imaging quality resulted from breathing artifact;
* without regularly follow-up information on recurrence location and time

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All T3 and T4 non-small cell lung cancers with surgery, and we retrospectively collected the preoperative enhanced chest CT and the recurrence location and time.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
disease free time and recurrence location | until the December 2023
  the time from the surgery time to the recurrence time

CONTACTS AND LOCATIONS:
Overall Officials: Guangming Lu, Study Director — Department of Radiology, Jinling Hospital
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang EH, Corso CD, Rutter CE, Park HS, Chen AB, Kim AW, Wilson LD, Decker RH, Yu JB. Postoperative Radiation Therapy Is Associated With Improved Overall Survival in Incompletely Resected Stage II and III Non-Small-Cell Lung Cancer. J Clin Oncol. 2015 Sep 1;33(25):2727-34. doi: 10.1200/JCO.2015.61.1517. Epub 2015 Jun 22. PMID 26101240
- [Background] Gillies RJ, Kinahan PE, Hricak H. Radiomics: Images Are More than Pictures, They Are Data. Radiology. 2016 Feb;278(2):563-77. doi: 10.1148/radiol.2015151169. Epub 2015 Nov 18. PMID 26579733
- [Background] Huang Y, Liu Z, He L, Chen X, Pan D, Ma Z, Liang C, Tian J, Liang C. Radiomics Signature: A Potential Biomarker for the Prediction of Disease-Free Survival in Early-Stage (I or II) Non-Small Cell Lung Cancer. Radiology. 2016 Dec;281(3):947-957. doi: 10.1148/radiol.2016152234. Epub 2016 Jun 27. PMID 27347764
- [Background] Yang H, Wang L, Shao G, Dong B, Wang F, Wei Y, Li P, Chen H, Chen W, Zheng Y, He Y, Zhao Y, Du X, Sun X, Wang Z, Wang Y, Zhou X, Lai X, Feng W, Shen L, Qiu G, Ji Y, Chen J, Jiang Y, Liu J, Zeng J, Wang C, Zhao Q, Yang X, Hu X, Ma H, Chen Q, Chen M, Jiang H, Xu Y. A combined predictive model based on radiomics features and clinical factors for disease progression in early-stage non-small cell lung cancer treated with stereotactic ablative radiotherapy. Front Oncol. 2022 Aug 2;12:967360. doi: 10.3389/fonc.2022.967360. eCollection 2022. PMID 35982975
- [Background] She Y, He B, Wang F, Zhong Y, Wang T, Liu Z, Yang M, Yu B, Deng J, Sun X, Wu C, Hou L, Zhu Y, Yang Y, Hu H, Dong D, Chen C, Tian J. Deep learning for predicting major pathological response to neoadjuvant chemoimmunotherapy in non-small cell lung cancer: A multicentre study. EBioMedicine. 2022 Dec;86:104364. doi: 10.1016/j.ebiom.2022.104364. Epub 2022 Nov 14. PMID 36395737
- [Background] Sawabata N, Matsumura A, Ohota M, Maeda H, Hirano H, Nakagawa K, Matsuda H; Thoracic Surgery Study Group of Osaka University. Cytologically malignant margins of wedge resected stage I non-small cell lung cancer. Ann Thorac Surg. 2002 Dec;74(6):1953-7. doi: 10.1016/s0003-4975(02)03993-0. PMID 12643379
- [Background] Akinci D'Antonoli T, Farchione A, Lenkowicz J, Chiappetta M, Cicchetti G, Martino A, Ottavianelli A, Manfredi R, Margaritora S, Bonomo L, Valentini V, Larici AR. CT Radiomics Signature of Tumor and Peritumoral Lung Parenchyma to Predict Nonsmall Cell Lung Cancer Postsurgical Recurrence Risk. Acad Radiol. 2020 Apr;27(4):497-507. doi: 10.1016/j.acra.2019.05.019. Epub 2019 Jul 6. PMID 31285150
- [Result] Ohguri T, Yahara K, Moon SD, Yamaguchi S, Imada H, Hanagiri T, Tanaka F, Terashima H, Korogi Y. Postoperative radiotherapy for incompletely resected non-small cell lung cancer: clinical outcomes and prognostic value of the histological subtype. J Radiat Res. 2012;53(2):319-25. doi: 10.1269/jrr.11082. Epub 2012 Feb 13. PMID 22327172
- [Result] Hancock JG, Rosen JE, Antonicelli A, Moreno A, Kim AW, Detterbeck FC, Boffa DJ. Impact of adjuvant treatment for microscopic residual disease after non-small cell lung cancer surgery. Ann Thorac Surg. 2015 Feb;99(2):406-13. doi: 10.1016/j.athoracsur.2014.09.033. Epub 2014 Dec 17. PMID 25528723
- [Result] Sawabata N, Maeda H, Matsumura A, Ohta M, Okumura M; Thoracic Surgery Study Group of Osaka University. Clinical implications of the margin cytology findings and margin/tumor size ratio in patients who underwent pulmonary excision for peripheral non-small cell lung cancer. Surg Today. 2012 Feb;42(3):238-44. doi: 10.1007/s00595-011-0031-6. Epub 2011 Nov 10. PMID 22072149
- [Result] Qi LL, Wang JW, Yang L, Huang Y, Zhao SJ, Tang W, Jin YJ, Zhang ZW, Zhou Z, Yu YZ, Wang YZ, Wu N. Natural history of pathologically confirmed pulmonary subsolid nodules with deep learning-assisted nodule segmentation. Eur Radiol. 2021 Jun;31(6):3884-3897. doi: 10.1007/s00330-020-07450-z. Epub 2020 Nov 21. PMID 33219848
- [Result] Kelsey CR, Marks LB, Hollis D, Hubbs JL, Ready NE, D'Amico TA, Boyd JA. Local recurrence after surgery for early stage lung cancer: an 11-year experience with 975 patients. Cancer. 2009 Nov 15;115(22):5218-27. doi: 10.1002/cncr.24625. PMID 19672942
- [Result] Zwanenburg A, Vallieres M, Abdalah MA, Aerts HJWL, Andrearczyk V, Apte A, Ashrafinia S, Bakas S, Beukinga RJ, Boellaard R, Bogowicz M, Boldrini L, Buvat I, Cook GJR, Davatzikos C, Depeursinge A, Desseroit MC, Dinapoli N, Dinh CV, Echegaray S, El Naqa I, Fedorov AY, Gatta R, Gillies RJ, Goh V, Gotz M, Guckenberger M, Ha SM, Hatt M, Isensee F, Lambin P, Leger S, Leijenaar RTH, Lenkowicz J, Lippert F, Losnegard A, Maier-Hein KH, Morin O, Muller H, Napel S, Nioche C, Orlhac F, Pati S, Pfaehler EAG, Rahmim A, Rao AUK, Scherer J, Siddique MM, Sijtsema NM, Socarras Fernandez J, Spezi E, Steenbakkers RJHM, Tanadini-Lang S, Thorwarth D, Troost EGC, Upadhaya T, Valentini V, van Dijk LV, van Griethuysen J, van Velden FHP, Whybra P, Richter C, Lock S. The Image Biomarker Standardization Initiative: Standardized Quantitative Radiomics for High-Throughput Image-based Phenotyping. Radiology. 2020 May;295(2):328-338. doi: 10.1148/radiol.2020191145. Epub 2020 Mar 10. PMID 32154773